CLINICAL TRIAL: NCT02724787
Title: CAP - Using Emotion Regulation to Decrease Aggression in Veterans With PTSD
Brief Title: Using Emotion Regulation to Decrease Aggression in Veterans With PTSD
Acronym: (EMDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLE-001-W14; W81XWH-12-PHTBI-CA (Other Grant/Funding Number: VA Clincial Science Research and Development)
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Post-Traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Veterans; Aggression; Emotion regulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Trial (Other): All Veterans will receive the same emotion regulation treatment titled, Manage Emotions to Reduce Aggression.
  Interventions: Behavioral: Manage Emotions to Reduce Aggression (MERA)

INTERVENTIONS:
Behavioral: Manage Emotions to Reduce Aggression (MERA) — MERA is a 3-session group treatment that teaches Veterans the purpose of emotions, how trauma and combat can increase emotions, and how to better regulate them. The skills use cognitive-behavioral and mindfulness techniques to help Veteran better regulate their emotions. These skills are commonly used in clinical practice, but have not been delivered in 3 sessions.

SUMMARY:
Impulsive aggression (IA) is common among Veterans with posttraumatic stress disorder (PTSD), and PTSD is one of the most prevalent post deployment mental health conditions affecting Afghanistan and Iraq Veterans. An inability to manage one's emotions (emotion dysregulation) is an underlying mechanism of IA. Reducing IA and increasing use of PTSD evidence-based psychotherapies are two critical missions for the Veterans Health Administration.

This research supports these missions by providing a 3-session emotion regulation training (Manage Emotions to Reduce Aggression) to Veterans in order to teach them how to manage emotions and prepare for PTSD treatment. This is an open trail, so all Veterans who meet the inclusion criteria will be allowed to receive the treatment. Each Veteran's level of aggression and emotion dysregulation will be measured at the beginning and end to the treatment. By enhancing Veterans' abilities to cope with trauma-related emotions and feel equipped to initiate PTSD treatments, this research aims to help Veterans decrease IA and ultimately recover from PTSD.

DETAILED DESCRIPTION:
In this pilot study for the Consortium to Alleviate PTSD, Shannon Miles, PhD, of the James A. Haley Veterans' Hospital in Tampa, Florida, and her study team will work with post-9/11 combat Veterans with PTSD and impulsive aggression. The Veterans will be identified as having impulsive aggression if they report having engaged in at least three episodes of aggression within the past month. The investigators will provide training in emotion regulation via an innovative three-session training called Managing Emotions to Reduce Aggression, or MERA.

The goal of the pilot study is to test the feasibility of MERA in reducing impulsive aggression. A secondary goal is to prepare Veterans for psychotherapy for PTSD. One reason that too few Veterans seek PTSD treatment may be that they fear that they will not be able to control their emotional responses when they begin treatment. The investigators for this study believe that equipping Veterans with emotion regulation skills and knowledge about PTSD treatments may help them initiate, complete, and benefit from evidence-based psychotherapies.

MERA is provided in a three-session, condensed time frame to make it accessible to Veterans whose careers, school, and families compete with treatment time. The training is delivered in a group format and incorporates emotion education, cognitive-behavioral and acceptance-based skills training, and information about what emotional experiences to expect from PTSD treatments. Study participants will undergo weekly assessments for emotion regulation and aggression. Following the MERA training, study participants will be followed by CAP investigators to monitor whether they seek out, receive, and complete evidence-based psychotherapies for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male Veteran who served in Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF)/Operation New Dawn (OND)
* Currently meets criteria for a PTSD diagnosis, determined by the Clinician-Administered PTSD Scale-5
* Engaged in at least 3 self-reported impulsive aggression acts in the last month, measured by the Overt Aggression Scale.58:

  * yelling
  * throwing objects
  * hitting objects/people in the last month
* Impulsive aggression is his/her primary form of aggression, determined by having a higher Impulsive Aggression subscore than a Premeditated Aggression subscore on the Impulsive Premeditated Aggression Scale
* Because aggressors are poor historians when reporting their aggression frequency, each Veteran must agree to allow an independent aggression rater (live-in partner, family member, or roommate) verify the number of aggressive acts, using the Overt Aggression Scale
* No psychotropic medication change for six weeks prior to the assessment and agreement not to ask for a medication change for the duration of the study

Exclusion Criteria:

Veterans who meet the following criteria will be excluded:

* Previously began Prolonged Exposure (PE) or Cognitive Processing Therapy (CPT)
* Is currently suicidal with intent of self-harm in the last week
* Is currently homicidal with plans to hurt a specific person
* Is unable to complete self-report measures
* Does not have an independent aggression rater
* Has severe alcohol consumption patterns (Alcohol Use Disorders Identification Test), severe drug use consumption patterns (Drug Use Disorders Identification Test), active psychosis, or mania (MINI)
* Had a psychotropic medication change within 6 weeks prior to the pretraining assessment. Veterans receiving general mental health services or non- PE or CPT psychotherapy will be allowed to participate in this study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon R. Miles, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: CAP - Using Emotion Regulation to Decrease Aggression in Veterans with PTSD — https://tango.uthscsa.edu/strongstar/subs/cpinfo.asp?prj=506

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Trial
Started | 24
Completed | 22 (22 completed treatment. 20 participants returned for post-treatment assessment.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Trial
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.17 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported ethnicity
  Participants
    Hispanic or Latino | 5
    Not Hispanic or Latino | 19
    Unknown or Not Reported | 0
Number of Overt Aggression Scale [Mean (Standard Deviation); unit: events] — Frequency count of aggressive acts in the past week. Theoretical minimum score = 0; no limit on maximum value. Higher values = greater frequency of aggression
  events | 30.79 (24.0)
Difficulties in Emotion Regulation [Mean (Standard Deviation); unit: units on a scale] — Total score was used in this study. Theoretical minimum value = 36; theoretical maximum value = 180. Higher scores indicate worse emotion regulation.
  units on a scale | 117.92 (19.1)
Emotion Regulation Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The ERQ is a self report measure with 2 factors that assess specific emotion regulation strategies: cognitive reappraisal (6 items; changing the way one thinks about a situation) and expressive suppression (4 items; not expressing the emotion outwardly but feeling it internally). More effective emotion regulation is indicated by higher cognitive reappraisal scores and lower expressive suppression scores. Cognitive reappraisal theoretical minimum score = 6; maximum score = 42. Expressive Suppression theoretical minimum score = 4; maximum score = 28.
  units on a scale
    Suppression Subscale | 17.42 (4.75)
    Cognitive Reappraisal Subscale | 25.42 (7.71)

OUTCOME MEASURES:

1. Primary Outcome: Overt Aggression Scale
Description: The Overt Aggression Scale (OAS) is a 17-item self-report measure that assesses frequency of different aggression acts, including verbal and physical aggression against self, other, and objects. Theoretical minimum score = 0; there is no bounded maximum value. Higher values = greater frequency of aggression.
Time Frame: Given 3 weeks after last MERA session. Assess aggressive events in past week.
Population: 22 participants completed the treatment. 20 participants returned for the post-treatment assessment.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Open Trial
Number analyzed (Participants) | 20
events | 14.2 (11.40)

2. Primary Outcome: Total Score Difficulties in Emotion Regulation Scale
Description: The Difficulties in Emotion Regulation Scale (DERS) is a 36- item self-report measure with 6 different emotion-dysregulation factors: nonacceptance of emotional responses, difficulties engaging in goal-directed behaviors, impulse-control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Total score was used in this study. Theoretical minimum value = 36; theoretical maximum value = 180. Higher scores indicate worse emotion regulation.
Time Frame: Given 3 weeks after last MERA session. Assess emotion dysregulation in past month.
Population: 22 participants completed the treatment. 20 participants returned for the post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 20
score on a scale | 107.45 (19.51)

3. Primary Outcome: Emotion Regulation Questionnaire
Description: ERQ is a 10-item self-report measure with 2 factors that assess specific emotion regulation strategies: cognitive reappraisal (6 items; changing the way one thinks about a situation) and expressive suppression (4 items; not expressing the emotion outwardly but feeling it internally). More effective emotion regulation is indicated by higher cognitive reappraisal scores and lower expressive suppression scores. Theoretical minimum score for cognitive reappraisal = 6; theoretical maximum score = 42. Theoretical minimum score for expressive suppression = 4; theoretical maximum score = 28.
Time Frame: Given 3 weeks after last MERA session. Assess emotion regulation strategies used in past week.
Population: 22 participants completed the treatment. 20 participants returned for the post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 20
score on a scale
  Suppression Subscale | 16.85 (3.44)
  Cognitive Reappraisal | 26.55 (5.83)

4. Primary Outcome: Exit Interview - Ratings of Therapist and Treatment
Description: The exit interview was created by the study team and has 3 questions that asks: 1.) how understanding the therapist was, 2.) how helpful the therapist was in learning skills, and 3.) how helpful MERA was in managing emotions.
  Scale for all questions:
  * 1 = Not at all understanding / helpful
  * 2 = A little bit understanding / helpful
  * 3 = Moderately understanding / helpful
  * 4 = Very understanding / helpful Higher scores reflect greater understanding or helpfulness.
Time Frame: Given 3 weeks after last MERA session.
Population: 22 participants completed the treatment. 20 participants returned for the post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 20
score on a scale
  How understanding therapist was | 3.94 (0.24)
  How helpful therapist was | 3.68 (0.75)
  How helpful MERA was | 3.15 (0.88)

5. Primary Outcome: Exit Interview - Use of Skills
Description: The exit interview was created by the study team and has 8 questions that asks: 1.) "Are you using _____skill?". Scores = percentage of the sample that was using the skill during the week before the post treatment assessment. Percentages could range from 0% to 100% of the sample. Higher scores represent more of the sample using the skill.
Time Frame: Given 3 weeks after last MERA session. Assess emotion regulation strategies used in past week.
Population: 22 participants completed the treatment. 20 participants returned for the post-treatment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Trial
Number analyzed (Participants) | 20
Participants
  Controlled breathing | 17
  Remember values | 14
  Grounding | 14
  Realistic thoughts | 14
  Progressive muscle relaxation | 12
  Visualization | 12
  Recognizing emotions | 12
  Increasing positive emotions | 7

ADVERSE EVENTS:
Time Frame: AE data were collected after the consent form was signed until the post-treatment assessment, an average of 10 weeks.
Description: We considered any clinically significant deterioration in physical, psychological, mental, cognitive, or psychosocial health status of the subject as a change from baseline as an AE. We did not use specific Adverse Event Terms.
Arm/Group | Open Trial
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Trial (N=24)
Hospitalization (Blood and lymphatic system disorders) | 1 — Diagnosed with cancer
Increase in symptoms (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT02724787/Prot_SAP_000.pdf